CLINICAL TRIAL: NCT03828266
Title: Abdominal Infectious Complications After Gastrointestinal Surgery in China: a Multi-centered Prospective Registry
Brief Title: Prediction of Abdominal Complications After GastroEnterological Surgery
Acronym: PACAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Ziyu Li, MD, Prof. Dr., Peking University
Other Study IDs: 2018YJZ56
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Complication; Anastomotic Leak; Gastrointestinal Cancer
MeSH Terms: conditions — Anastomotic Leak; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Patients will undergo routine clinical practice. There is no additional intervention.

SUMMARY:
The aim of this multi-centered study is to understand the epidemiology of infectious complications after gastrointestinal surgery in China. In total, 17 centers from China will prospectively register their patients undergo gastric or colorectal surgeries. Patient demographic data, operation information, and postoperative data including the infectious complications and the outcomes will be registered. We expect to include 2000 gastric and 2000 colorectal patients within one year and the study is expected to be finished in 2020.

DETAILED DESCRIPTION:
All participating hospital will log in on a website based e-CRF system. Researchers need to register the patient information that three time-points: admission, after surgery, after discharge.

The detailed registered information includes:

I. Basic and surgical information:

Age, height, weight, history of abdominal surgery, ASA score, surgical procedure, extent of lymph node dissection, extent of resection, time of surgery, amount of bleeding, whether it is emergency surgery, whether it is combined with organ resection, whether it is palliative resection, whether combined with preoperative treatment, whether combined with preoperative infection and intraoperative complications.

II. Postoperative information:

Primary lesion histological type, margin, pathological stage (pTNM); other complications, postoperative death and discharge time, CRP, PCT, WBC levels.

III. Abdominal Infection information:

Abdominal infection (Y/N), anastomotic leakage (Y/N), intervention, outcome.

ELIGIBILITY:
Inclusion Criteria:

* Planned gastrointestinal surgery.
* Inform consent received.

Exclusion Criteria:

* Endoscopic surgery.
* Inform consent denied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergo gastrointestinal (GI) surgery for GI tumor.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Abdominal Infection rate after gastrectomy. | From surgery until discharge, up to 90 days.
  Abdominal Infection includes anastomotic leakage and other intra-abdominal infectious complications.
Abdominal Infection rate after colorectal surgery. | From surgery until discharge, up to 90 days.
  Abdominal Infection includes anastomotic leakage and other intra-abdominal infectious complications.

SECONDARY OUTCOMES:
Classification of Abdominal Infection after Surgery | From surgery until discharge, up to 90 days.
  Severity classification scored based on Clavien-Dindo score, it includes five different scales indicating different severity of the complication.
Diagnosis time of Abdominal Complication | From surgery until discharge, up to 90 days.
  1-3 days after surgery; 4-7 days after surgery; >1wk after surgery
Outcome of Abdominal Infection Treatment | From surgery until discharge, up to 90 days.
  Cured before discharge, not cured before discharge, death.

CONTACTS AND LOCATIONS:
Overall Officials: Ziyu Li, MD PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (19):
- China (19):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Xiamen University First Hospital, Xiamen, Fujian
  - Guangdong People's Hospital, Guangzhou, Guangdong
  - The First Affilliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - South Hospital, Guanzhou, Guangdong
  - Nanchang University First Hospital, Nanchang, Jiangxi
  - Jilin University Second Hospital, Changchun, Jilin
  - Dalian Medical University First Hospital, Dalian, Liaoning
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - Shandong Provincial Hospital, Jinan, Shandong
  - Qingdao University Affiliated Hospital, Qingdao, Shandong
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Xi'an Jiao Tong University First Hospital, Xi’an, Shanxi
  - Hangzhou First Hospital, Hangzhou, Zhejiang
  - Run Run Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu Z, Gu T, Wang X, Wei T, Shan F, Li Z, Ji J; PACAGE study group. Surgical quality and health utilization of gastric cancer surgery in China: a post hoc analysis of the Prevalence of Abdominal Complications After Gastroenterological Surgery study. BMJ Surg Interv Health Technol. 2025 Jul 15;7(1):e000332. doi: 10.1136/bmjsit-2024-000332. eCollection 2025. PMID 40671863